CLINICAL TRIAL: NCT01998360
Title: Rapid, Minimally-invasive Voluntary Adult Male Circumcision: a Quasi-experimental Study
Brief Title: Rapid, Minimally-invasive Voluntary Adult Male Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simunye Primary Health Care (Other)
Responsible Party: Principal Investigator, Peter Millard, PI, Simunye Primary Health Care
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Unicirc 002
Record Dates: First submitted 2013-10-11; First posted 2013-11-28 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Circumcision
Keywords: Circumcision; Voluntary medical male circumcision; Minimally-invasive; HIV prevention
MeSH Terms: interventions — Tissue Adhesives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unicirc with tissue adhesive (Experimental): Excision of foreskin with Unicirc device and sealing wound with tissue adhesive
  Interventions: Procedure: Unicirc with tissue adhesive
- Surgical control (Active Comparator): Surgical circumcision using forceps guided, dorsal slit, or sleeve method
  Interventions: Procedure: Surgical Control

INTERVENTIONS:
Procedure: Surgical Control — The study is quasi-experimental, because the open surgical controls are not contemporaneous. They were performed at the same center as part of Unicirc 001 trial with the same conditions as the subsequent 50 Unicirc circumcisions.
  Arms: Surgical control
Procedure: Unicirc with tissue adhesive — Excision of foreskin with Unicirc device and wound sealing with tissue adhesive
  Arms: Unicirc with tissue adhesive

SUMMARY:
This study will evaluate a new, minimally-invasive surgical circumcision technique for men, which is easy to learn and perform, is safe, and is associated with high patient satisfaction and excellent cosmetic results.

DETAILED DESCRIPTION:
Voluntary medical male circumcision (VMMC) is a priority preventive intervention for HIV transmission. Currently, the most widely used VMMC technique in South Africa is open surgical circumcision.

According to the Framework for Clinical Evaluation of Devices for Adult Male Circumcision (WHO, 2011): "WHO and other health authorities wish to identify one or more devices that (a) would make the VMMC safer, easier, and quicker; (b) would have more rapid healing than current methods and/or might entail less risk of HIV transmission in the post-operative period; (c) could be performed safely by health-care providers with a minimal level of training; and (d) would be cost-effective compared to standard surgical methods for male circumcision scale up."

This quasi-experimental compares the open surgical technique to an alternative minimally-invasive technique using the disposable Unicirc device with tissue adhesive. The controls come from a separate randomized controlled trial (Unicirc 001) that was conducted just prior to the Unicirc 002 case series of 50 subjects. The investigators postulate that VMMC using the Unicirc device meets WHO criteria for the ideal method to scale up: it is an easier technique to learn and perform, requires less intraoperative time, is safer for both surgeons and patients, heals quicker, and is more cost effective than other currently available techniques. The disposable nature of the device is an immense advantage as it eliminates the need to sterilize and can therefore be used in resource-limited settings. It also reduces the chances of infection caused by contaminated instruments.

ELIGIBILITY:
Inclusion Criteria:

Healthy men at least 18 years of age requesting circumcision

No anatomical penile abnormalities or infections

Able to provide informed consent to participate

Willing to participate in follow-up visits -

Exclusion Criteria:

Current illness

Penile abnormality or infection which contraindicates or would complicate circumcision

History of bleeding disorder

Past reaction to local anesthetic

-

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Goldstuck, MB ChB, Study Director — Simunye Primary Health Care
Locations (1):
- Simunye Primary Healthcare, Mitchells Plain, Western Cape, South Africa

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unicirc With Tissue Adhesive | Surgical Control
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unicirc With Tissue Adhesive | Surgical Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Duration
Description: The number of minutes required to perform the surgical procedure
Time Frame: 1 hour
Measure: Median (Inter-Quartile Range); unit: Min
Arm/Group | Unicirc With Tissue Adhesive | Surgical Control
Number analyzed (Participants) | 50 | 50
Min | 9.0 [8.5 to 10.0] | 22.6 [18.4 to 27.0]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Bleeding, hematoma, infection and other rare adverse events
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | Unicirc With Tissue Adhesive | Surgical Control
Number analyzed (Participants) | 50 | 50
participants | 4 | 9

3. Secondary Outcome: Blood Loss
Description: Number of ml of blood lost during the procedure, as assessed by the surgeon
Time Frame: During procedure (up to 1 hour)
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Unicirc With Tissue Adhesive | Surgical Control
Number analyzed (Participants) | 50 | 50
ml | 1.5 [1.5 to 1.5] | 5.5 [5.5 to 12]

4. Secondary Outcome: Number of Participants With Complete Epithelialization (Completely Healed) at 4 Weeks
Description: The number of participants with complete epithelialization (completely healed) at 4 weeks
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | Unicirc With Tissue Adhesive | Surgical Control
Number analyzed (Participants) | 50 | 50
participants | 49 | 49

5. Secondary Outcome: Cosmetic Result
Description: Regular: scar line straight without any irregularity
  Irregular: Some irregularity to scar line
  Scalloped: wavy appearane to scar line
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Unicirc With Tissue Adhesive | Surgical Control
Number analyzed (Participants) | 50 | 50
participants
  Regular | 50 | 20
  Irregular | 0 | 8
  Scalloped | 0 | 22

ADVERSE EVENTS:
Arm/Group | Unicirc With Tissue Adhesive | Surgical Control
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 4/50 | 9/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unicirc With Tissue Adhesive (N=50) | Surgical Control (N=50)
Post-op bleeding or hematoma (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Post-op infection (Infections and infestations) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No